CLINICAL TRIAL: NCT00201240
Title: A Phase 2 Single Arm Trial of HLA-Matched Transplants, CD34+ Enriched, T-Cell Depleted Peripheral Blood Stem Cells Isolated by CliniMACS System in the Treatment of Patients With AML in 1st or 2nd Morphologic Complete Remission (BMTCTN0303)
Brief Title: Acute Myeloid Leukemia T Cell Depletion to Improve Transplants in Adults With Acute Myeloid Leukemia (BMT CTN 0303)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0303; U01HL069254 (NIH); U01HL069249 (NIH); U01HL069278 (NIH); U01HL069294 (NIH); U01HL069315 (NIH); U01HL069348 (NIH); 284 (Other: NHLBI)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2017-08

CONDITIONS: Leukemia, Myelocytic, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD34+ selection with CliniMACS device (Experimental): T cell depletion using Miltenyi device
  Interventions: Biological: CD34+ selection with CliniMACS device

INTERVENTIONS:
Biological: CD34+ selection with CliniMACS device — CD34+ cell selection will be performed according to procedures given in the CliniMACS Users Operating Manual and institutional Standard Operating Procedures (SOPs) in place and validated at the study sites. CliniMACS (Miltenyi device) to target CD34+ >5 x 10*6/kg and CD3+ < 1 x 10*5/kg
  Other Names: T Cell Depletion

SUMMARY:
This study is a single arm Phase II, multicenter trial. It is designed to determine whether the anticipated endpoints for a T cell depleted transplant arm of a planned prospective randomized trial comparing T cell depleted and unmodified hematopoietic allografts are likely to be achieved in a multicenter study conducted by the Blood and Marrow Transplant Clinical Trials Network (BMT CTN or Network). The study population is patients with acute myeloid leukemia (AML) in first or second morphologic complete remission. The enrollment is 45 patients.

Based on published results of unmodified transplants from HLA-matched siblings applied to patients with AML in first or second morphologic complete remission, a significant improvement in results with a graft modified as specified in this protocol would be expected if disease-free survival (DFS) at 6 months was greater than 75%, the true incidence of transplant-related mortality at 1 year was less than 30%, and the DFS rate at 2 years was greater 70% for patients transplanted in first remission and less than 60% for patients transplanted in second remission. Additional secondary endpoints include the following: graft failure rate and incidences of acute grade II-IV and chronic graft-versus-host disease (GVHD). Additionally, the trial will have target specific doses of CD34+ progenitors and CD3+ T cells to be obtained following fractionation with the CliniMACS system. Based on the results of this trial, a Phase III trial comparing T cell depleted peripheral blood stem cell transplants (PBSCT) with unmanipulated bone marrow or unmanipulated PBSCT will be designed.

DETAILED DESCRIPTION:
BACKGROUND:

Allogeneic hematopoietic cell transplantation is an accepted therapy for AML. Transplants of unmodified HLA-matched related bone marrow or peripheral blood stem cells following conditioning with total body irradiation (TBI) and cyclophosphamide or VP-16 or busulfan and cyclophosphamide have led to sustained DFS rates of 45-60% for adults transplanted in first complete remission (CR1) and 40-53% for patients transplanted in second complete remission (CR2). In several single center and multicenter cooperative group prospective trials comparing HLA-matched allogeneic transplants to chemotherapy in the treatment of AML in CR1, DFS rates for the transplant arm were almost invariably superior; however, these advantages were statistically significant in only a minority of the cooperative group studies conducted. In each study, the risk of relapse was significantly lower for patients receiving allogeneic transplants. However, this advantage was counterbalanced by transplant-related mortality, principally reflecting infections complicating GVHD and its treatment.

DESIGN NARRATIVE:

Despite increased risks of infection, development of effective T cell depletion (TCD) techniques for prevention of GVHD and tolerable modifications of regimens for pre-transplant cytoreduction that secure consistent engraftment offer the potential for significant decreases in transplant-related mortality. Furthermore, the use of TCD transplants in the treatment of patients with AML is not associated with substantial increases in the incidence of relapse. Several single center trials indicate highly encouraging long-term results, particularly for patients with AML in CR1 or CR2. Although the number of cases in each single center series is limited, the consistency of the results suggests that the use of an effective technique for TCD together with an adequate cytoreductive regimen might yield transplant results superior to those achieved with unmodified grafts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML with or without prior history of myelodysplastic syndrome based on the World Health Organization criteria at the following stages:

  * First morphologic complete remission (CR)
  * Second morphologic CR
* If prior history of central nervous system (CNS) involvement, no evidence of active CNS leukemia during the pre-transplant evaluation (no evidence of leukemic blasts in cerebrospinal fluid)
* First or second CR was achieved after no more than two cycles of induction (or re-induction for patients in second CR) chemotherapy
* No more than 6 months elapsed from documentation of CR to transplant for patients in first CR, or 3 months for patients in second CR.
* A 6/6 HLA antigen (A, B, DRB1)-compatible sibling donor; the match may be determined at serologic level for HLA-A and HLA-B loci; DRB1 must be matched at least at low-resolution using DNA typing techniques; HLA-C will be typed at the serologic level, but not included in the match algorithm
* Karnofsky performance status greater than 70%
* Life expectancy greater than 8 weeks
* Diffusing capacity of the lung for carbon monoxide (DLCO) of at least 40% (corrected for hemoglobin) with no symptomatic pulmonary disease
* Left ventricular ejection fraction (LVEF) by Multi Gated Acquisition Scan (MUGA) or echocardiogram greater than 40%
* Serum creatinine greater than 2 mg/dL, bilirubin greater than 2 mg/dL, and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels at least 3 times the upper limit of normal at time of enrollment
* Willingness of both the patient and the donor to participate

Exclusion Criteria:

* M3-AML (acute promyelocytic leukemia) in first CR
* Acute leukemia following blast transformation of prior chronic myelogenous leukemia (CML) or other myeloproliferative disease
* M4Eo-AML with inv 16 in first CR
* AML with t(8;21) in first CR
* Participation in other clinical trials that involve investigational drugs or devices except with permission from the Medical Monitor
* Evidence of active Hepatitis B or C infection or evidence of cirrhosis
* HIV positive
* Uncontrolled diabetes mellitus
* If proven or probable invasive fungal infection, infection must be controlled; patients may be on prophylactic anti-fungal agents, but are not permitted to be on anti-fungal agents for therapeutic purposes (i.e., active treatment for disease)
* Uncontrolled viral or bacterial infection (currently taking medication without clinical improvement)
* Documented allergy to iron dextran or murine proteins
* Pregnant or breastfeeding; women of childbearing age must avoid becoming pregnant while in the study
* Prior autologous or allogeneic hematopoietic stem cell transplantation (HSCT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Devine, MD, Study Chair — Ohio State/Arthur G. James Cancer Hospital; Parameswaran Hari, MD, Principal Investigator — Medical College of Wisconsin; Hillard Lazarus, MD, Principal Investigator — University Hospitals of Cleveland/Case Western; Lloyd Damon, MD, Principal Investigator — University of California, San Francisco; Richard O'Reilly, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Robert Soiffer, MD, Principal Investigator — Dana Farber Cancer Institute/Brigham & Women's Hospital; Anthony Stein, MD, Principal Investigator — City of Hope National Medical Center; John DiPersio, MD, PhD, Principal Investigator — Washington University/Barnes Jewish Hospital; Edward Stadtmauer, MD, Principal Investigator — University of Pennsylvania
Locations (8):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Dana Farber Cancer Institute/Brigham & Women's Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Keever-Taylor CA, Devine SM, Soiffer RJ, Mendizabal A, Carter S, Pasquini MC, Hari PN, Stein A, Lazarus HM, Linker C, Goldstein SC, Stadtmauer EA, O'Reilly RJ. Characteristics of CliniMACS(R) System CD34-enriched T cell-depleted grafts in a multicenter trial for acute myeloid leukemia-Blood and Marrow Transplant Clinical Trials Network (BMT CTN) protocol 0303. Biol Blood Marrow Transplant. 2012 May;18(5):690-7. doi: 10.1016/j.bbmt.2011.08.017. Epub 2011 Aug 26. PMID 21875505
- [Result] Devine SM, Carter S, Soiffer RJ, Pasquini MC, Hari PN, Stein A, Lazarus HM, Linker C, Stadtmauer EA, Alyea EP 3rd, Keever-Taylor CA, O'Reilly RJ. Low risk of chronic graft-versus-host disease and relapse associated with T cell-depleted peripheral blood stem cell transplantation for acute myelogenous leukemia in first remission: results of the blood and marrow transplant clinical trials network protocol 0303. Biol Blood Marrow Transplant. 2011 Sep;17(9):1343-51. doi: 10.1016/j.bbmt.2011.02.002. Epub 2011 Feb 12. PMID 21320619
- [Result] Pasquini MC, Devine S, Mendizabal A, Baden LR, Wingard JR, Lazarus HM, Appelbaum FR, Keever-Taylor CA, Horowitz MM, Carter S, O'Reilly RJ, Soiffer RJ. Comparative outcomes of donor graft CD34+ selection and immune suppressive therapy as graft-versus-host disease prophylaxis for patients with acute myeloid leukemia in complete remission undergoing HLA-matched sibling allogeneic hematopoietic cell transplantation. J Clin Oncol. 2012 Sep 10;30(26):3194-201. doi: 10.1200/JCO.2012.41.7071. Epub 2012 Aug 6. PMID 22869882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from October2005 through December 2008
Groups:
- T Cell Depletion: T cell depletion using Miltenyi device for patients with acute myeloid leukemia (AML) in first or second complete remission
Period: Overall Study
Arm/Group | T Cell Depletion
Started | 47
Completed | 44
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- T Cell Depletion: T cell depletion using Miltenyi device for patients with AML in first or second complete remission
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
Age, Customized [Number; unit: participants] — Age of the participant in years
  participants
    <20 | 0
    20-29 | 7
    30-39 | 4
    40-49 | 14
    50-59 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 44
Karnofsky Performance Status [Number; unit: participants] — Karnofsky performance status of participants at baseline. The range is 0 to 100 with 100 being the best.
  participants
    100% | 17
    90% | 17
    80% | 8
    70% | 2
Leukemia stage [Number; unit: participants] — First complete remission (CR1) is achieved after an initial treatment. Second complete remission (CR2) is achieved after a second treatment when a relapse has occured. Complete remission (CR) is defined according to the revised recommendations of the international working group: Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, et al. Revised recommendations of the international working group for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in acute myeloid leukemia. J Clin Oncol 21(24): 4642-9, 2003.
  participants
    CR1 | 37
    CR2 | 7
Cytogenetic risk [Number; unit: participants]
  Favorable | 1
  Intermediate | 28
  Unfavorable | 14
  Unknown | 1
Recipient CMV Status [Number; unit: participants] — Cytomegalovirus (CMV)
  participants
    Positive | 17
    Negative | 27

OUTCOME MEASURES:

1. Primary Outcome: Probability of Disease-free Survival (DFS) at 6 Months Post-transplant (Death or Relapse Will be Considered Events for This Endpoint)
Description: The primary analysis will consist of estimating the 6-month DFS (from day of enrollment) probability based on the Kaplan-Meier product limit estimator. The 6-month DFS probability and confidence interval will be calculated. All registered patients will be considered for this analysis.
Time Frame: 6 months
Population: All transplanted patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of patients | 81.8 [70.3 to 93.4]

2. Secondary Outcome: Leukemia Relapse
Description: To assess the incidence of acute leukemia relapse from day of transplant, a cumulative incidence curve will be computed along with a 95% confidence interval. Death prior to relapse will be considered as a competing risk.
Time Frame: Months 12 and 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  12 months | 20.6 [8.4 to 32.8]
  36 months | 23.7 [10.5 to 37.0]

3. Secondary Outcome: Neutrophil Engraftment
Description: Time to neutrophil engraftment is measured by determining the first of three consecutive measurements of absolute neutrophil count ≥ 500/uL following conditioning regimen induced nadir, starting from Day 0.
Time Frame: 28 day
Measure: Median (Full Range); unit: days
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
days | 12 [9 to 19]

4. Secondary Outcome: Platelet Engraftment
Description: Time to platelet engraftment is measured by determining the first of three consecutive measurements of platelet count ≥ 20,000/uL without platelet transfusion support for seven days, starting from Day 0.
Time Frame: 6 Months
Measure: Median (Full Range); unit: days
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
days | 16 [13 to 159]

5. Secondary Outcome: Graft Failure
Description: Primary graft failure is defined as the failure to achieve an ANC > 500 cells/µL by Day +30. Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in neutrophil counts < 500 cells/µL, unresponsive to growth factor therapy.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
participants
  Primary Graft Failure | 0
  Secondary Graft Failure | 1

6. Secondary Outcome: Acute Graft Versus Host Disease (GVHD)
Description: Incidence and severity of acute GVHD will be graded according to the BMT CTN MOP.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  Grades II - IV | 22.7 [10.2 to 35.3]
  Grades III - IV | 4.5 [0 to 10.8]

7. Secondary Outcome: Chronic Graft Versus Host Disease (GVHD)
Description: Incidence and severity of chronic GVHD will be scored according to the BMT CTN MOP.
Time Frame: Year 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  Limited/extensive | 19.0 [6.8 to 31.1]
  Extensive only | 6.8 [0 to 14.4]

8. Secondary Outcome: Transplant Related Mortality
Description: Death occurring in a patient in continuing complete remission.
Time Frame: Months 12, 24, and 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  12 months | 14 [3.4 to 24]
  24 months | 20 [7.1 to 32.7]
  36 months | 23.2 [9.3 to 37.1]

9. Secondary Outcome: Determination of Infusional Toxicity
Time Frame: 28 day
Population: No data collected
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 0

10. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the minimum time interval of times to relapse/recurrence, to death or to the last follow-up, from the time of transplant.
Time Frame: Months 6, 12, and 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  6 months | 81.8 [70.3 to 93.4]
  12 months | 66 [52 to 80]
  36 months | 53 [37 to 69]

11. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from transplant to death or last follow-up.
Time Frame: Months 12 and 36
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
percentage of participants
  12 months | 77 [65 to 90]
  36 months | 56 [40 to 73]

12. Secondary Outcome: CD34+ and CD3+ Cell Doses
Description: Total CD34+ and CD3+ cell doses will be calculated based on results of flow cytometric analysis.
Time Frame: Day 0
Measure: Median (Full Range); unit: cells per kilogram
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
cells per kilogram
  CD34+ (x10^6) | 7.9 [2.4 to 31.3]
  CD3+ (x10^3) | 6.6 [1.1 to 84.9]

13. Secondary Outcome: Post-transplant Lymphoproliferative Disorder (PTLD)
Description: PTLD is defined as increased Epstein Barr Virus viremia requiring clinical intervention.
Time Frame: Year 2
Measure: Number; unit: participants
Arm/Group | T Cell Depletion
Number analyzed (Participants) | 44
participants | 8

ADVERSE EVENTS:
Arm/Group | T Cell Depletion
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2006-11-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT00201240/Prot_SAP_ICF_000.pdf